CLINICAL TRIAL: NCT03329235
Title: Intraosseous With Intra-articular Injection of Platelet Rich Plasma Versus Hyaluronic Acid in Treatment of Knee Osteoarthritis
Brief Title: Intraosseous With Intra-articular Injection of Platelet Rich Plasma in Treatment of Knee Osteoarthritis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cangzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cangzhou Central Hospital
Record Dates: First submitted 2017-03-03; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intraosseous and intra-articular (Experimental): injection of PRP 2 ml
  Interventions: Drug: PRP
- intra-articular PRP (Active Comparator): injection PRP 2 ml
  Interventions: Drug: PRP
- Intra-articular injection of HA (Active Comparator): injection of HA 2 ml
  Interventions: Drug: HA

INTERVENTIONS:
Drug: PRP — platelet rich plasma
  Arms: Intraosseous and intra-articular; intra-articular PRP
Drug: HA — hyaluronic acid
  Arms: Intra-articular injection of HA

SUMMARY:
The aim of this study was to compare the efficacy of treatment in three groups of patients with knee osteoarthritis (OA) given a combination of intraosseous with intra-articular injection of platelet rich plasma (PRP), intra-articular injection of PRP and a single application of hyaluronic acid (HA).

DETAILED DESCRIPTION:
Methods Eighty-six patients from January 2015 to June 2015 with grade II to grade III knee osteoarthritis according to the Kellgren-Lawrence classification were randomly divided into 3 groups to receive either PRP or HA. Group A received intra-articular injection of PRP 2 ml combination with medial tibial plateau and medial femoral condyle injection of PRP 2 ml (once more 2 weeks later). Group B were treated with 2 ml of PRP intra-articular injection every 14 days for a total of two injections. Group C received intra-articular injection of hyaluronic acid 2 ml every 7 days for five injections. All patients were evaluated by the Visual Analogue Scale (VAS) and the Western Ontario and McMaster Universities (WOMAC) score before the treatment and at 1st, 3rd, 6th, 12th and 18th months.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral symptomatic knee with pain for at least 1 month or swelling.
* Radiographic findings of knee degeneration (Kellgren-Lawrence score of II - III).
* Age 40-73 years.
* Body mass index (BMI) 18-32.5).
* Knee stability without a severe trauma history.

Exclusion Criteria:

* Bilateral knee osteoarthritis indicative of treatment for both knees.
* Kellgren-Lawrence score greater than III.
* BMI >32.
* Age >73 years.
* Systemic autoimmune rheumatic diseases and blood disorders.
* Active immunosuppressive or anticoagulant therapy.
* Intra-articular injection to the knee within the previous 1 year or previous joint infection.
* use of corticosteroids for 3 weeks before the procedure.
* use of nonsteroidal anti-inflammatory drugs (NSAIDs) in the 3 weeks before treatment.

Ages: 40 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
WOMAC scores | At the 18th month
  The evaluation was performed with WOMAC, which were recorded on a five-point Likert scale scoring, with a response of "none" scored as 0, "mild" as 1, "moderate" as 2, "severe" as 3 and "extreme" as 4.

IPD SHARING:
Plan to Share IPD: Yes